CLINICAL TRIAL: NCT04252586
Title: An Open-label Extension Trial to Investigate the Long-term Safety of Cannabidiol Oral Solution (GWP42003-P, CBD-OS) in Patients With Rett Syndrome
Brief Title: A Long-term Safety Study of Cannabidiol Oral Solution (GWP42003-P, CBD-OS) in Patients With Rett Syndrome
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was terminated due to COVID-19 pandemic and recruitment challenges in the parent study (GWND18064 - NCT03848832).
Sponsor: Jazz Pharmaceuticals (Industry)
Collaborators: GW Pharmaceuticals Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GWND19002; 2019-001605-24 (EudraCT Number)
Record Dates: First submitted 2020-01-30; First posted 2020-02-05 (Actual); Results first posted 2022-08-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-07

CONDITIONS: Rett Syndrome; RTT
Keywords: Cannabidiol; CBD; Epidiolex; GWP42003-P
MeSH Terms: conditions — Rett Syndrome | interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GWP42003-P (Experimental): 100 milligrams per milliliter (mg/mL) GWP42003-P oral solution, taken twice daily (morning and evening).
  Interventions: Drug: GWP42003-P

INTERVENTIONS:
Drug: GWP42003-P — GWP42003-P presented as an oral solution containing cannabidiol in the excipients sesame oil with anhydrous ethanol, sweetener (sucralose), and strawberry flavoring
  Other Names: Cannabidiol; CBD; Epidiolex; CBD-OS

SUMMARY:
This study will be conducted to evaluate the long-term safety of cannabidiol oral solution (GWP42003-P, CBD-OS) in participants with Rett syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Participant has completed all scheduled visits of the treatment phase of the randomized controlled trial (RCT), GWND18064 (NCT03848832), and has transitioned to open-label extension (OLE) by the point of RCT follow-up
* Participant (if possessing adequate understanding, in the investigator's opinion) and/or the participant(s)/legal representative is willing and able to give informed consent/assent for participation in the trial.
* Participant and the participant's caregiver are willing and able (in the investigator's opinion) to comply with all trial requirements (including the completion of all caregiver assessments by the same caregiver throughout the trial).
* Ability to swallow the investigational medicinal product (IMP) provided as a liquid solution, or the ability for the IMP to be delivered via gastrostomy (G) or nasogastric (NG) feeding tube (only G- or NG-tubes made from polyurethane or silicon are allowed).
* Participant and/or parent(s)/legal representative is willing to allow the responsible authorities to be notified of participation in the trial, if mandated by local law.
* Participant and/or parent(s)/legal representative is willing to allow the participant's primary care practitioner (if the participant has one) and consultant (if the participant has one) to be notified of participation in the trial, if the primary care practitioner/consultant is different from the investigator.

Exclusion Criteria:

* Participant meets the withdrawal criteria (including clinically significant abnormal laboratory values), in the investigator's opinion.
* Participant met during the RCT the criteria for permanent IMP discontinuation (unless in the case of an adverse event [AE], if the AE was not considered related with the IMP; participants that met alanine aminotransferase (ALT)/aspartate aminotransferase (AST) elevations discontinuation criteria must be excluded).
* Females of childbearing potential, unless willing to ensure that they or their partner use a highly effective method of birth control (e.g., combined [estrogen and progestogen containing] hormonal contraception associated with inhibition of ovulation [oral, intravaginal, or transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, or implantable], intrauterine devices/hormone-releasing systems, bilateral tubal occlusion, vasectomized partner, sexual abstinence during the trial and for 3 months after the last dose
* Participant has been previously enrolled and dosed in this trial.
* Participant is unwilling to abstain from donation of blood during the trial.
* Male participants who are fertile (i.e., after puberty unless permanently sterile by bilateral orchidectomy) and with a partner of childbearing potential unless agree to ensure that they use male contraception (e.g., condom) or remain sexually abstinent during the trial and for 3 months after the last dose

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (31):
- United States (14):
  - Clinical Trial Site, Birmingham, Alabama
  - Clinical Trial Site, La Jolla, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Saint Paul, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, The Bronx, New York
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Greenwood, South Carolina
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Houston, Texas
- Australia (2):
  - Clinical Trial Site, Perth
  - Clinical Trial Site, South Brisbane
- Canada (2):
  - Clinical Trial Site, Toronto
  - Clinical Trial Site, Vancouver
- Italy (5):
  - Clinical Trial Site, Genova
  - Clinical Trial Site, Messina
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Rome
  - Clinical Trial Site, Siena
- Spain (5):
  - Clinical Trial Site #1, Barcelona
  - Clinical Trial Site #2, Barcelona
  - Clinical Trial Site #1, Madrid
  - Clinical Trial Site #2, Madrid
  - Clinical Trial Site, Valencia
- United Kingdom (3):
  - Clinical Trial Site, Edinburgh
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 21 participants who had previously participated in the randomized, double-blind, placebo-controlled trial GWND18064 (NCT03848832) entered this open label extension study.
Groups:
- GWP42003-P: Participants who received oral GWP42003-P (5 mg/kg/day) on Day 1. After 1 week, depending on clinical response and tolerability, the participants' dose may have been increased at the Investigator's discretion to weekly increments of 5 mg/kg/day up to 15 mg/kg/day GWP42003-P. Participants remained on a stable dose of GWP42003-P for the duration of the maintenance period of the trial (up to 104 weeks), with the option for doses to be decreased or increased to a maximum dose of 20 mg/kg/day based on clinical response and tolerability, as deemed necessary by the Investigator.
Period: Overall Study
Arm/Group | GWP42003-P
Started | 21
Completed | 0
Not Completed | 21
Not completed — Withdrawal by parent/guardian | 3
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Study terminated by sponsor | 4
Not completed — Sponsor request | 10
Not completed — Did not complete treatment period | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were assessed in the Safety Analysis Set which was defined as all participants who received at least one dose of GWP42003-P in the study.
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.2 (5.59)
Age, Customized [Count of Participants; unit: Participants]
  2-5 years | 6
  6-12 years | 9
  13-19 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (TEAEs), Discontinuations Due to AEs, Serious AEs, and Treatment-related AEs
Description: Adverse events (AEs) were defined as any new unfavorable/unintended signs/symptoms (including abnormal laboratory findings when relevant) or diagnosis or worsening of a pre-existing condition that occurs during the study. TEAEs were defined as the AEs that started or worsened in severity or seriousness following the first dose of GWP42003-P. A serious AE was defined as any AE that results in any of the following outcomes: death, life-threatening adverse experience, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or cancer, any other experience that suggests a significant hazard, contraindication, side effect or precaution that may require medical or surgical intervention to prevent one of the outcomes listed above, or an event that changes the risk/benefit ratio of the study.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 16 (Day 767) in the OLE
Population: Adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Any TEAE | 19
  Treatment-related TEAEs | 7
  TEAEs leading to discontinuation | 3
  Treatment-related TEAE leading to discontinuation | 1
  Serious TEAEs | 5
  Treatment-related serious TEAEs | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Clinical Laboratory Parameters From the Baseline at Any Time Post-dose
Description: Treatment-emergent clinical parameters were defined as the following: Treatment-emergent alanine transferase (ALT) > 3×upper limit of normal (ULN), > 5×ULN and > 8×ULN; Treatment-emergent aspartate aminotransferase (AST) > 3×ULN, > 5×ULN and > 8×ULN; Treatment-emergent ALT or AST > 3×ULN, > 5×ULN and > 8×ULN; Treatment-emergent ALT or AST > 3×ULN and either bilirubin > 2×ULN or international normalized ratio (INR) > 1.5.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Clinical laboratory parameters were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- GWP42003-P: Participants received GWP42003-P (5 mg/kg/day]) for 1 week. Depending on clinical response and tolerability, the participants' dose was increased in weekly increments of 5 mg/kg/day up to 15 mg/kg/day GWP42003-P. Participant remained on a stable dose of GWP42003-P for the duration of the maintenance period of the trial (up to 104 weeks), with the option for doses to be decreased or increased to a maximum dose of 20 mg/kg/day based on clinical response and tolerability, as deemed necessary by the investigator.
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Treatment-emergent ALT >3xULN | 1
  Treatment-emergent ALT >5xULN | 0
  Treatment-emergent ALT >8xULN | 0
  Treatment-emergent AST >3xULN | 0
  Treatment-emergent AST >5xULN | 0
  Treatment-emergent AST >8xULN | 0
  Treatment-emergent ALT or AST >3xULN | 1
  Treatment-emergent ALT or AST >5xULN | 0
  Treatment-emergent ALT or AST >8xULN | 0
  Treatment-emergent ALT or AST > 3×ULN and either bilirubin > 2×ULN or INR > 1.5 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Changes in Vital Sign Values of Blood Pressure From the Baseline at Any Time Post-dose
Description: Potentially clinically significant vital sign values of blood pressure (BP) were defined as sitting systolic BP (mmHg) change: < -20 or > 20 mmHg and sitting diastolic BP change: < -10 or > 10 mmHg. Vital sign measurements were taken in a sitting position at rest for 5 minutes. Blood pressure readings were recorded using the same arm throughout the trial, when possible.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 15 (Day 739) in the OLE
Population: Vital signs were assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Systolic BP Change <-20 mmHg, Baseline | 4
  Systolic BP Change <-20 mmHg, Day 29: number analyzed (Participants) | 20
  Systolic BP Change <-20 mmHg, Day 29 | 2
  Systolic BP Change <-20 mmHg, Day 57: number analyzed (Participants) | 18
  Systolic BP Change <-20 mmHg, Day 57 | 1
  Systolic BP Change <-20 mmHg, Day 85: number analyzed (Participants) | 19
  Systolic BP Change <-20 mmHg, Day 85 | 1
  Systolic BP Change <-20 mmHg, Day 141: number analyzed (Participants) | 14
  Systolic BP Change <-20 mmHg, Day 141 | 2
  Systolic BP Change <-20 mmHg, Day 197: number analyzed (Participants) | 9
  Systolic BP Change <-20 mmHg, Day 197 | 2
  Systolic BP Change <-20 mmHg, Day 281: number analyzed (Participants) | 2
  Systolic BP Change <-20 mmHg, Day 281 | 0
  Systolic BP Change <-20 mmHg, Day 365: number analyzed (Participants) | 2
  Systolic BP Change <-20 mmHg, Day 365 | 0
  Systolic BP Change <-20 mmHg, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Systolic BP Change <-20 mmHg, End of Treatment (up to Day 729) | 1
  Systolic BP Change <-20 mmHg, Day 739: number analyzed (Participants) | 3
  Systolic BP Change <-20 mmHg, Day 739 | 1
  Systolic BP Change >20 mmHg, Baseline | 1
  Systolic BP Change >20 mmHg, Day 29: number analyzed (Participants) | 20
  Systolic BP Change >20 mmHg, Day 29 | 1
  Systolic BP Change >20 mmHg, Day 57: number analyzed (Participants) | 18
  Systolic BP Change >20 mmHg, Day 57 | 3
  Systolic BP Change >20 mmHg, Day 85: number analyzed (Participants) | 19
  Systolic BP Change >20 mmHg, Day 85 | 2
  Systolic BP Change >20 mmHg, Day 141: number analyzed (Participants) | 14
  Systolic BP Change >20 mmHg, Day 141 | 0
  Systolic BP Change >20 mmHg, Day 197: number analyzed (Participants) | 9
  Systolic BP Change >20 mmHg, Day 197 | 0
  Systolic BP Change >20 mmHg, Day 281: number analyzed (Participants) | 2
  Systolic BP Change >20 mmHg, Day 281 | 0
  Systolic BP Change >20 mmHg, Day 365: number analyzed (Participants) | 2
  Systolic BP Change >20 mmHg, Day 365 | 0
  Systolic BP Change >20 mmHg, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Systolic BP Change >20 mmHg, End of Treatment (up to Day 729) | 2
  Systolic BP Change >20 mmHg, Day 739: number analyzed (Participants) | 3
  Systolic BP Change >20 mmHg, Day 739 | 0
  Diastolic BP Change <-10 mmHg, Baseline | 7
  Diastolic BP Change <-10 mmHg, Day 29: number analyzed (Participants) | 20
  Diastolic BP Change <-10 mmHg, Day 29 | 4
  Diastolic BP Change <-10 mmHg, Day 57: number analyzed (Participants) | 18
  Diastolic BP Change <-10 mmHg, Day 57 | 4
  Diastolic BP Change <-10 mmHg, Day 85: number analyzed (Participants) | 19
  Diastolic BP Change <-10 mmHg, Day 85 | 2
  Diastolic BP Change <-10 mmHg, Day 141: number analyzed (Participants) | 14
  Diastolic BP Change <-10 mmHg, Day 141 | 3
  Diastolic BP Change <-10 mmHg, Day 197: number analyzed (Participants) | 9
  Diastolic BP Change <-10 mmHg, Day 197 | 3
  Diastolic BP Change <-10 mmHg, Day 281: number analyzed (Participants) | 2
  Diastolic BP Change <-10 mmHg, Day 281 | 0
  Diastolic BP Change <-10 mmHg, Day 365: number analyzed (Participants) | 2
  Diastolic BP Change <-10 mmHg, Day 365 | 0
  Diastolic BP Change <-10 mmHg, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Diastolic BP Change <-10 mmHg, End of Treatment (up to Day 729) | 3
  Diastolic BP Change <-10 mmHg, Day 739: number analyzed (Participants) | 3
  Diastolic BP Change <-10 mmHg, Day 739 | 0
  Diastolic BP Change >10 mmHg, Baseline | 4
  Diastolic BP Change >10 mmHg, Day 29: number analyzed (Participants) | 20
  Diastolic BP Change >10 mmHg, Day 29 | 9
  Diastolic BP Change >10 mmHg, Day 57: number analyzed (Participants) | 18
  Diastolic BP Change >10 mmHg, Day 57 | 4
  Diastolic BP Change >10 mmHg, Day 85: number analyzed (Participants) | 19
  Diastolic BP Change >10 mmHg, Day 85 | 4
  Diastolic BP Change >10 mmHg, Day 141: number analyzed (Participants) | 14
  Diastolic BP Change >10 mmHg, Day 141 | 3
  Diastolic BP Change >10 mmHg, Day 197: number analyzed (Participants) | 9
  Diastolic BP Change >10 mmHg, Day 197 | 1
  Diastolic BP Change >10 mmHg, Day 281: number analyzed (Participants) | 2
  Diastolic BP Change >10 mmHg, Day 281 | 0
  Diastolic BP Change >10 mmHg, Day 365: number analyzed (Participants) | 2
  Diastolic BP Change >10 mmHg, Day 365 | 0
  Diastolic BP Change >10 mmHg, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Diastolic BP Change >10 mmHg, End of Treatment (up to Day 729) | 5
  Diastolic BP Change >10 mmHg, Day 739: number analyzed (Participants) | 3
  Diastolic BP Change >10 mmHg, Day 739 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in the Vital Sign Values of Pulse Rate From the Baseline at Any Time Post-dose
Description: Potentially clinically significant vital sign values of pulse rate were defined as pulse rate change: < -10 or > 10 beats per minute. Vital sign measurements were taken in a sitting position at rest for 5 minutes.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 15 (Day 739) in the OLE
Population: Pulse rate was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Pulse Rate Change <-10beats/min, Baseline | 9
  Pulse Rate Change <-10beats/min, Day 29: number analyzed (Participants) | 20
  Pulse Rate Change <-10beats/min, Day 29 | 8
  Pulse Rate Change <-10beats/min, Day 57: number analyzed (Participants) | 18
  Pulse Rate Change <-10beats/min, Day 57 | 7
  Pulse Rate Change <-10beats/min, Day 85: number analyzed (Participants) | 19
  Pulse Rate Change <-10beats/min, Day 85 | 7
  Pulse Rate Change <-10beats/min, Day 141: number analyzed (Participants) | 14
  Pulse Rate Change <-10beats/min, Day 141 | 2
  Pulse Rate Change <-10beats/min, Day 197: number analyzed (Participants) | 9
  Pulse Rate Change <-10beats/min, Day 197 | 5
  Pulse Rate Change <-10beats/min, Day 281: number analyzed (Participants) | 2
  Pulse Rate Change <-10beats/min, Day 281 | 1
  Pulse Rate Change <-10beats/min, Day 365: number analyzed (Participants) | 2
  Pulse Rate Change <-10beats/min, Day 365 | 1
  Pulse Rate Change <-10beats/min, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Pulse Rate Change <-10beats/min, End of Treatment (up to Day 729) | 6
  Pulse Rate Change <-10beats/min, Day 739: number analyzed (Participants) | 3
  Pulse Rate Change <-10beats/min, Day 739 | 0
  Pulse Rate Change >10beats/min, Baseline | 5
  Pulse Rate Change >10beats/min, Day 29: number analyzed (Participants) | 20
  Pulse Rate Change >10beats/min, Day 29 | 2
  Pulse Rate Change >10beats/min, Day 57: number analyzed (Participants) | 18
  Pulse Rate Change >10beats/min, Day 57 | 3
  Pulse Rate Change >10beats/min, Day 85: number analyzed (Participants) | 19
  Pulse Rate Change >10beats/min, Day 85 | 3
  Pulse Rate Change >10beats/min, Day 141: number analyzed (Participants) | 14
  Pulse Rate Change >10beats/min, Day 141 | 3
  Pulse Rate Change >10beats/min, Day 197: number analyzed (Participants) | 9
  Pulse Rate Change >10beats/min, Day 197 | 1
  Pulse Rate Change >10beats/min, Day 281: number analyzed (Participants) | 2
  Pulse Rate Change >10beats/min, Day 281 | 0
  Pulse Rate Change >10beats/min, Day 365: number analyzed (Participants) | 2
  Pulse Rate Change >10beats/min, Day 365 | 0
  Pulse Rate Change >10beats/min, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Pulse Rate Change >10beats/min, End of Treatment (up to Day 729) | 4
  Pulse Rate Change >10beats/min, Day 739: number analyzed (Participants) | 3
  Pulse Rate Change >10beats/min, Day 739 | 2

5. Primary Outcome: Number of Participants With Clinically Significant Percent Change in Body Weight From the Baseline at Any Time Post-dose
Description: Clinically significant body weight changes were defined as the percent change in body weight (≤7% change or ≥7% change).
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Body weight was assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Weight Percent Change ≤7%, Baseline | 1
  Weight Percent Change ≤7%, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Weight Percent Change ≤7%, End of Treatment (up to Day 729) | 1
  Weight Percent Change ≥7%, Baseline | 8
  Weight Percent Change ≥7%, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Weight Percent Change ≥7%, End of Treatment (up to Day 729) | 10

6. Primary Outcome: Number of Participants With At Least One Post Open Label Extension Baseline Flagged ECG Result
Description: Electrocardiogram assessments were performed for QTcB and QTcF >450 msec, >480 msec, and >500 msec. QTcB = corrected QT interval with Bazette correction. QTcF = QTc corrected by Fridericia.
Time Frame: Visit 4 (Day 29) up to Visit 15 (Day 739) in the OLE
Population: Electrocardiogram assessments were performed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 20
Participants
  QTcB Interval, Aggregate > 450 msec, Day 29 | 4
  QTcB Interval, Aggregate > 450 msec, Day 57: number analyzed (Participants) | 18
  QTcB Interval, Aggregate > 450 msec, Day 57 | 0
  QTcB Interval, Aggregate > 450 msec, Day 85: number analyzed (Participants) | 19
  QTcB Interval, Aggregate > 450 msec, Day 85 | 4
  QTcB Interval, Aggregate > 450 msec, Day 141: number analyzed (Participants) | 14
  QTcB Interval, Aggregate > 450 msec, Day 141 | 0
  QTcB Interval, Aggregate > 450 msec, Day 197: number analyzed (Participants) | 9
  QTcB Interval, Aggregate > 450 msec, Day 197 | 0
  QTcB Interval, Aggregate > 450 msec, Day 365: number analyzed (Participants) | 2
  QTcB Interval, Aggregate > 450 msec, Day 365 | 0
  QTcB Interval, Aggregate > 450 msec, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  QTcB Interval, Aggregate > 450 msec, End of Treatment (up to Day 729) | 4
  QTcB Interval, Aggregate > 450 msec, Day 739: number analyzed (Participants) | 3
  QTcB Interval, Aggregate > 450 msec, Day 739 | 0
  QTcB Interval, Aggregate > 480 msec, Day 29 | 0
  QTcB Interval, Aggregate > 480 msec, Day 57: number analyzed (Participants) | 18
  QTcB Interval, Aggregate > 480 msec, Day 57 | 0
  QTcB Interval, Aggregate > 480 msec, Day 85: number analyzed (Participants) | 19
  QTcB Interval, Aggregate > 480 msec, Day 85 | 1
  QTcB Interval, Aggregate > 480 msec, Day 141: number analyzed (Participants) | 14
  QTcB Interval, Aggregate > 480 msec, Day 141 | 0
  QTcB Interval, Aggregate > 480 msec, Day 197: number analyzed (Participants) | 9
  QTcB Interval, Aggregate > 480 msec, Day 197 | 0
  QTcB Interval, Aggregate > 480 msec, Day 365: number analyzed (Participants) | 2
  QTcB Interval, Aggregate > 480 msec, Day 365 | 0
  QTcB Interval, Aggregate > 480 msec, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  QTcB Interval, Aggregate > 480 msec, End of Treatment (up to Day 729) | 1
  QTcB Interval, Aggregate > 480 msec, Day 739: number analyzed (Participants) | 3
  QTcB Interval, Aggregate > 480 msec, Day 739 | 0
  QTcB Interval, Aggregate > 500 msec, Day 29 | 0
  QTcB Interval, Aggregate > 500 msec, Day 57: number analyzed (Participants) | 18
  QTcB Interval, Aggregate > 500 msec, Day 57 | 0
  QTcB Interval, Aggregate > 500 msec, Day 85: number analyzed (Participants) | 19
  QTcB Interval, Aggregate > 500 msec, Day 85 | 0
  QTcB Interval, Aggregate > 500 msec, Day 141: number analyzed (Participants) | 14
  QTcB Interval, Aggregate > 500 msec, Day 141 | 0
  QTcB Interval, Aggregate > 500 msec, Day 197: number analyzed (Participants) | 9
  QTcB Interval, Aggregate > 500 msec, Day 197 | 0
  QTcB Interval, Aggregate > 500 msec, Day 365: number analyzed (Participants) | 2
  QTcB Interval, Aggregate > 500 msec, Day 365 | 0
  QTcB Interval, Aggregate > 500 msec, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  QTcB Interval, Aggregate > 500 msec, End of Treatment (up to Day 729) | 0
  QTcB Interval, Aggregate > 500 msec, Day 739: number analyzed (Participants) | 3
  QTcB Interval, Aggregate > 500 msec, Day 739 | 0
  QTcF Interval, Aggregate > 450 msec, Day 29 | 0
  QTcF Interval, Aggregate > 450 msec, Day 57: number analyzed (Participants) | 18
  QTcF Interval, Aggregate > 450 msec, Day 57 | 0
  QTcF Interval, Aggregate > 450 msec, Day 85: number analyzed (Participants) | 19
  QTcF Interval, Aggregate > 450 msec, Day 85 | 1
  QTcF Interval, Aggregate > 450 msec, Day 141: number analyzed (Participants) | 14
  QTcF Interval, Aggregate > 450 msec, Day 141 | 0
  QTcF Interval, Aggregate > 450 msec, Day 197: number analyzed (Participants) | 9
  QTcF Interval, Aggregate > 450 msec, Day 197 | 0
  QTcF Interval, Aggregate > 450 msec, Day 365: number analyzed (Participants) | 2
  QTcF Interval, Aggregate > 450 msec, Day 365 | 0
  QTcF Interval, Aggregate > 450 msec, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  QTcF Interval, Aggregate > 450 msec, End of Treatment (up to Day 729) | 0
  QTcF Interval, Aggregate > 450 msec, Day 739: number analyzed (Participants) | 3
  QTcF Interval, Aggregate > 450 msec, Day 739 | 0
  QTcF Interval, Aggregate > 480 msec, Day 29 | 0
  QTcF Interval, Aggregate > 480 msec, Day 57: number analyzed (Participants) | 18
  QTcF Interval, Aggregate > 480 msec, Day 57 | 0
  QTcF Interval, Aggregate > 480 msec, Day 85: number analyzed (Participants) | 19
  QTcF Interval, Aggregate > 480 msec, Day 85 | 0
  QTcF Interval, Aggregate > 480 msec, Day 141: number analyzed (Participants) | 14
  QTcF Interval, Aggregate > 480 msec, Day 141 | 0
  QTcF Interval, Aggregate > 480 msec, Day 197: number analyzed (Participants) | 9
  QTcF Interval, Aggregate > 480 msec, Day 197 | 0
  QTcF Interval, Aggregate > 480 msec, Day 365: number analyzed (Participants) | 2
  QTcF Interval, Aggregate > 480 msec, Day 365 | 0
  QTcF Interval, Aggregate > 480 msec, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  QTcF Interval, Aggregate > 480 msec, End of Treatment (up to Day 729) | 0
  QTcF Interval, Aggregate > 480 msec, Day 739: number analyzed (Participants) | 3
  QTcF Interval, Aggregate > 480 msec, Day 739 | 0
  QTcF Interval, Aggregate > 500 msec, Day 29 | 0
  QTcF Interval, Aggregate > 500 msec, Day 57: number analyzed (Participants) | 18
  QTcF Interval, Aggregate > 500 msec, Day 57 | 0
  QTcF Interval, Aggregate > 500 msec, Day 85: number analyzed (Participants) | 19
  QTcF Interval, Aggregate > 500 msec, Day 85 | 0
  QTcF Interval, Aggregate > 500 msec, Day 141: number analyzed (Participants) | 14
  QTcF Interval, Aggregate > 500 msec, Day 141 | 0
  QTcF Interval, Aggregate > 500 msec, Day 197: number analyzed (Participants) | 9
  QTcF Interval, Aggregate > 500 msec, Day 197 | 0
  QTcF Interval, Aggregate > 500 msec, Day 365: number analyzed (Participants) | 2
  QTcF Interval, Aggregate > 500 msec, Day 365 | 0
  QTcF Interval, Aggregate > 500 msec, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  QTcF Interval, Aggregate > 500 msec, End of Treatment (up to Day 729) | 0
  QTcF Interval, Aggregate > 500 msec, Day 739: number analyzed (Participants) | 3
  QTcF Interval, Aggregate > 500 msec, Day 739 | 0

7. Primary Outcome: Number of Participants With Any Changes In Menstruation Cycle at Any Time Post-dose
Description: Participants were evaluated for any changes to typical menstrual cycles, duration of menstrual cycles, and typical strength of the menstrual cycles during the study.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Changes in menstruation cycle was assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Any change to typical cycle, Yes; Day 1 | 1
  Any change to typical cycle, No; Day 1 | 1
  Any change to typical cycle; Day 1 Unknown/Missing | 19
  Typical duration of menstruation cycle, <3 days; Day 1 | 0
  Typical duration of menstruation cycle, 3-7 days; Day 1 | 1
  Typical duration of menstruation cycle, >7 days; Day 1 | 0
  Typical duration of menstruation cycle; Day 1 Unknown/Missing | 20
  Typical strength of menstruation cycle, Light; Day 1 | 1
  Typical strength of menstruation cycle, Moderate; Day 1 | 0
  Typical strength of menstruation cycle, Heavy; Day 1 | 0
  Typical strength of menstruation cycle, Other; Day 1 | 0
  Typical strength of menstruation cycle; Day 1 Unknown/Missing | 20
  Any change to typical cycle, Yes; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Any change to typical cycle, Yes; End of Treatment (up to Day 729) | 3
  Any change to typical cycle, No; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Any change to typical cycle, No; End of Treatment (up to Day 729) | 3
  Any change to typical cycle; End of Treatment (up to Day 729) Unknown/Missing: number analyzed (Participants) | 18
  Any change to typical cycle; End of Treatment (up to Day 729) Unknown/Missing | 12
  Typical duration of menstruation cycle, <3 days; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical duration of menstruation cycle, <3 days; End of Treatment (up to Day 729) | 0
  Typical duration of menstruation cycle, 3-7 days; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical duration of menstruation cycle, 3-7 days; End of Treatment (up to Day 729) | 3
  Typical duration of menstruation cycle, >7 days; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical duration of menstruation cycle, >7 days; End of Treatment (up to Day 729) | 0
  Typical duration of menstruation cycle; End of Treatment (up to Day 729) Unknown/Missing: number analyzed (Participants) | 18
  Typical duration of menstruation cycle; End of Treatment (up to Day 729) Unknown/Missing | 15
  Typical strength of menstruation cycle, Light; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical strength of menstruation cycle, Light; End of Treatment (up to Day 729) | 1
  Typical strength of menstruation cycle, Heavy; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical strength of menstruation cycle, Heavy; End of Treatment (up to Day 729) | 2
  Typical strength of menstruation cycle, Moderate; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical strength of menstruation cycle, Moderate; End of Treatment (up to Day 729) | 0
  Typical strength of menstruation cycle, Other; End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Typical strength of menstruation cycle, Other; End of Treatment (up to Day 729) | 0
  Typical strength of menstruation cycle; End of Treatment (up to Day 729) Unknown/Missing: number analyzed (Participants) | 18
  Typical strength of menstruation cycle; End of Treatment (up to Day 729) Unknown/Missing | 15

8. Primary Outcome: Number of Participants With Suicidal Ideation or Behavior at the Baseline and at Any Time Post-dose
Description: Suicidal ideation and behavior was assessed by the investigator via a clinical interview with the caregiver. The questionnaire included following questions: Has the child expressed any wish to be dead?, Has the child made any suicide attempts?, Has the child shown any non-suicidal self-injurious behavior? The responses were recorded as Yes/No.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Suicidal ideation or behavior was assessed in participants with available data in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Has the child expressed any wish to be dead? Yes, Baseline | 0
  Has the child expressed any wish to be dead? No, Baseline | 16
  Has the child expressed any wish to be dead? Unknown/Missing, Baseline | 5
  Has the child expressed any wish to be dead? Yes, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Has the child expressed any wish to be dead? Yes, End of Treatment (up to Day 729) | 0
  Has the child expressed any wish to be dead? No, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Has the child expressed any wish to be dead? No, End of Treatment (up to Day 729) | 18
  Has the child made any suicide attempts? Yes, Baseline | 0
  Has the child made any suicide attempts? No, Baseline | 16
  Has the child made any suicide attempts? Unknown/Missing, Baseline | 5
  Has the child made any suicide attempts? Yes, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Has the child made any suicide attempts? Yes, End of Treatment (up to Day 729) | 0
  Has the child made any suicide attempts? No, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Has the child made any suicide attempts? No, End of Treatment (up to Day 729) | 18
  Has the child shown any non-suicidal self-injurious behavior? Yes, Baseline | 0
  Has the child shown any non-suicidal self-injurious behavior? Yes, usual behavior, Baseline | 3
  Has the child shown any non-suicidal self-injurious behavior? Yes, worsening behavior, Baseline | 0
  Has the child shown any non-suicidal self-injurious behavior? No, Baseline | 13
  Has the child shown any non-suicidal self-injurious behavior? Unknown/Missing, Baseline | 5
  Has the child shown any non-suicidal self-injurious behavior? Yes, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Has the child shown any non-suicidal self-injurious behavior? Yes, End of Treatment (up to Day 729) | 0
  Has child shown any non-suicidal self-injurious behavior? Yes, usual behavior, EOT (up to Day 729): number analyzed (Participants) | 18
  Has child shown any non-suicidal self-injurious behavior? Yes, usual behavior, EOT (up to Day 729) | 4
  Has child shown any non-suicidal self-injurious behavior? Yes, worse behavior, EOT (up to Day 729): number analyzed (Participants) | 18
  Has child shown any non-suicidal self-injurious behavior? Yes, worse behavior, EOT (up to Day 729) | 0
  Has child shown any non-suicidal self-injurious behavior? No, End of Treatment (up to Day 729): number analyzed (Participants) | 18
  Has child shown any non-suicidal self-injurious behavior? No, End of Treatment (up to Day 729) | 14

9. Primary Outcome: Mean Change From Baseline in Insulin-like Growth Factor-1 (IGF-1) Levels at End of Treatment
Description: Blood samples were collected to assess changes in serum IGF-1 levels. A negative mean change from baseline indicates a reduction in IGF-1 levels.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: IGF-1 levels were assessed in participants with available data in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P
Number analyzed (Participants) | 11
units on a scale | -41.1 (100.77)

10. Primary Outcome: Number of Participants With Changes in Tanner Staging at the Baseline and at End of Treatment
Description: Pubic hair growth and breast development of all adolescents were assessed by the investigator or caregiver using Tanner Staging categorization from 1 to 5.
  Stage 1- No glandular tissue; areola follows skin contours of chest; No pubic hair Stage 2- Breast bud forms; areola begins to widen; a small amount of long, downy hair with slight pigmentation on labia majora Stage 3- Breast begins to become more elevated and extends beyond borders of the areola, which continues to widen but remains in contour with surrounding breast; Hair becomes more coarse and curly and begins to extend laterally Stage 4- Increased breast size and elevation; areola and papilla form a secondary mound projecting from the contour of the surrounding breast; Adult-like hair quality, extending across pubis but sparing medial thighs Stage 5- Breast reaches final adult size; areola returns to the contour of the surrounding breast, with a projecting central papilla; Hair extends to medial surface of the thigh.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Changes in Tanner staging was assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
Participants
  Baseline, Tanner Stage 1 | 6
  Baseline, Tanner Stage 2 | 3
  Baseline, Tanner Stage 3 | 1
  Baseline, Tanner Stage 4 | 2
  Baseline, Tanner Stage 5 | 4
  Baseline, Tanner Stage Missing | 5
  End of Treatment (up to Day 729), Tanner Stage 1: number analyzed (Participants) | 18
  End of Treatment (up to Day 729), Tanner Stage 1 | 4
  End of Treatment (up to Day 729), Tanner Stage 2: number analyzed (Participants) | 18
  End of Treatment (up to Day 729), Tanner Stage 2 | 2
  End of Treatment (up to Day 729), Tanner Stage 3: number analyzed (Participants) | 18
  End of Treatment (up to Day 729), Tanner Stage 3 | 1
  End of Treatment (up to Day 729), Tanner Stage 4: number analyzed (Participants) | 18
  End of Treatment (up to Day 729), Tanner Stage 4 | 3
  End of Treatment (up to Day 729), Tanner Stage 5: number analyzed (Participants) | 18
  End of Treatment (up to Day 729), Tanner Stage 5 | 3
  End of Treatment (up to Day 729), Tanner Stage Missing: number analyzed (Participants) | 18
  End of Treatment (up to Day 729), Tanner Stage Missing | 5

11. Secondary Outcome: Mean Change From Baseline in Rett Syndrome Behaviour Questionnaire (RSBQ) Overall Score at End of Treatment
Description: RSBQ is a caregiver-completed questionnaire that assesses the overall condition (45 items) in individuals with Rett Syndrome. Each item is rated on a 3-point scale (0-2); 0 indicating an item that is "not true as far as you know," 1 indicating an item is "somewhat or sometimes true," and 2 indicating an item that is "very true or often true". " Item 31 ("Uses eye gaze to convey feelings, needs and wishes") is reverse-scored (0 indicating "very true or often true", 1 indicating "somewhat or sometimes true," and 2 indicating "not true as far as you know"). The total summed score ranges from 0 to 90, with higher scores representing greater severity. A negative mean change from baseline indicates an improvement in overall condition.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Rett Syndrome Behaviour Questionnaire (RSBQ) was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
units on a scale | -7.4 (14.93)

12. Secondary Outcome: Mean Clinical Global Impressions-Improvement (CGI-I) Continuous Score at End of Treatment
Description: CGI-I is a 7-point scale that requires the clinician to assess whether a patient's condition has improved or worsened relative to a baseline state at the beginning of the intervention. This was rated as: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; or 7 = very much worse. The mean continuous CGI-I score (averaged from each treatment enrolled under protocol and under annex) at Visit 14 (Day 729) is being reported. Higher mean scores indicate worse condition.
Time Frame: Visit 14 (Day 729) in the OLE
Population: Clinical Global Impressions - Improvement was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
score on a scale | 3.3 (1.15)

13. Secondary Outcome: Mean Clinician Global Impressions - Severity Scale (CGI-S) Continuous Score at End of Treatment
Description: CGI-S is a 7-point scale that requires the clinician to rate the severity of the participant's illness at the time of assessment relative to the clinician's experience with participants who had the same diagnosis. This was rated as: 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 =severely ill; or 7 = extremely ill. The mean continuous CGI-S score (averaged from each treatment enrolled under protocol and under annex) at Visit 14 (Day 729) is being reported. Higher scores indicate more severe disease.
Time Frame: Visit 14 (Day 729) in the OLE
Population: Clinician Global Impressions - Severity was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
score on a scale | 4.3 (0.96)

14. Secondary Outcome: Mean Change From Baseline in Children's Sleep Habits Questionnaire (CSHQ) Total Score at End of Treatment
Description: CSHQ is a caregiver-completed sleep screening instrument designed for school-aged children; which includes 33 items within 8 subscales:bedtime resistance (score range 6-18), sleep onset delay (range 1-3), sleep duration (range 3-9), sleep anxiety (range 4-12), night wakings (range 3-9), parasomnias (range 7-21), sleep-disordered breathing (range 3-9), daytime sleepiness (range 8-24). The 33 items range from 1 to 3, where 3="usually" (≥5 times/week), 2="sometimes" (2-4 times/week), and 1="rarely" (≤1 time/week); for items 31 and 32, 3=fall asleep, 2=very sleepy, 1=not sleepy. A score of 3 indicates greater severity; however, 6 items (1-Goes to bed at same time; 3-Falls asleep in own bed; 26-Wakes by himself; 2-Falls asleep in 20 minutes; 10-Sleeps the right amount; 11-Sleeps same amount each day) are reverse scored. The total summed score ranges from 33 to 99, with higher scores indicating disturbed sleep behavior. A negative mean change from baseline indicates improvement in sleep.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Children's Sleep Habits Questionnaire (CSHQ) was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
units on a scale | -3.0 (6.87)

15. Secondary Outcome: Mean Change From Baseline in 9-item Motor Behavioral Assessment (MBA-9) Total Score at End of Treatment
Description: MBA-9 is derived from the full MBA scale (37 Rett syndrome symptoms) by selecting the items deemed amenable to change and which reflected areas of meaningful clinical change. The MBA-9 includes 9 items (Regression of motor skills; Poor eye/social contact; Lack of sustained interest; Does not reach for objects or people; Chewing difficulties; Speech disturbance; Hand clumsiness; Dystonia; and Hypertonia/rigidity). For each item, the severity of current symptoms is rated by the investigator on a 5-point numerical scale ranging from 0 to 4 with higher scores representing greater severity (0 = normal or never; 1 = mild or rare; 2 = moderate or occasional; 3 = marked or frequent; 4 = very severe or constant). Total MBA-9 score was calculated by summing the scores of 9 different subscale items. The total summed score ranges from 0 to 36, with higher scores representing greater severity. A negative mean change from baseline indicates improvement in behavior.
Time Frame: Baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 14 (Day 729) in the OLE
Population: Motor Behavioral Assessment (MBA-9) was assessed in the Safety Analysis Set.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GWP42003-P
Number analyzed (Participants) | 21
units on a scale | 0.7 (5.19)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline of randomized controlled trial (RCT) Visit 1 (Day 1) up to Visit 16 (Day 767) in the OLE.
Description: A treatment-emergent adverse event (TEAE) are defined as adverse events (AEs) that started or worsened in severity or seriousness following the first dose of GWP42003-P.
Arm/Group | GWP42003-P
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=21)
Rett Syndrome (Congenital, familial and genetic disorders) | 1
COVID-19 (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Postoperative wound infection (Infections and infestations) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Status epilepticus (Nervous system disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GWP42003-P (N=21)
Neutropenia (Blood and lymphatic system disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
Pyrexia (General disorders) | 4
Otitis media (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Mean cell volume increased (Investigations) | 2
Monocyte count decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Epilepsy (Nervous system disorders) | 2
Seizure (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 2
Bruxism (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rett syndrome (Congenital, familial and genetic disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2

LIMITATIONS AND CAVEATS:
This trial was terminated due to enrollment challenges and the COVID-19 pandemic. Due to early termination and participants withdrawal, the number of participants was small and the length of treatment was reduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There IS an agreement between the Principal Investigator and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.

DOCUMENTS (2):
  • Study Protocol (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/86/NCT04252586/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/86/NCT04252586/SAP_001.pdf